CLINICAL TRIAL: NCT03316937
Title: Comparison of the Effect of Teflon vs Non-Teflon Hand Scalers in the Maintenance of Peri-Implant Tissue: A Randomized Clinical Trial
Brief Title: Comparison of the Effect of Teflon vs Non-Teflon Hand Scalers in the Maintenance of Peri-Implant Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Dayna Roemermann, Principal Investigator - Periodontics Resident, University of Manitoba
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: B2017:124
Record Dates: First submitted 2017-10-17; First posted 2017-10-23 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Surface Roughness; Maintenance of Dental Implants; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: The buccal and lingual surface of the 23 participants' crowns will be randomly assigned to receive scaling and root planing with either Teflon scalers, or non-Teflon scalers after implant crown delivery. Each patient will act as their own control.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teflon Scaler (Experimental): The buccal and lingual surface of the 23 participants' crowns will be randomly assigned to receive scaling and root planing with either Teflon scalers, or non-Teflon scalers after implant crown delivery. Each patient will act as their own control.
  Interventions: Procedure: Types of scalers
- Non Teflon Scaler (Experimental): The buccal and lingual surface of the 23 participants' crowns will be randomly assigned to receive scaling and root planing with either Teflon scalers, or non-Teflon scalers after implant crown delivery. Each patient will act as their own control.
  Interventions: Procedure: Types of scalers

INTERVENTIONS:
Procedure: Types of scalers — Scaling

SUMMARY:
The buccal and lingual surface of the 23 participants' crowns will be randomly assigned to receive scaling and root planing with either Teflon scalers, or non-Teflon scalers after implant crown delivery. Each patient will act as their own control.

Patients will receive scaling and root planing at 3, 6, 9 and 12 months by a calibrated dental hygienist. All surfaces of the implant will be debrided for 1 minute using a transversal movement. Each patient will receive oral hygiene instructions by the hygienist at the end of each maintenance therapy appointment. The participants will be instructed to use a Modified Stillman brushing technique twice per day and cross shoe shine flossing motion once per day. Each patient will be provided with a three-month home care kit with dental aids. These aids will consist of toothpaste, a toothbrush and implant floss.

Measurements will be taken at 0, 3, 6, 9 and 12 months by a calibrated periodontal resident. The parameters assessed at the implant site and patient level will be modified plaque index (IPI) by Mombelli, modified gingival index (IBOP) by Mombelli, implant probing depths (PD) at six sites, presence of keratinized gingiva (KT), recession (REC), Full mouth plaque index (FPI) and Full mouth bleeding on probing (FBOP).

The Peri-implant Crevicular Fluid will be collected at 0, 3, and 12 months by isolating the implant site from saliva and introducing Periopaper strips into the buccal, mesial, distal and lingual sites of the implant sulcus for 30 seconds. The strips will be placed in a sealed Eppendorf tubes and transported by portable freezer to the laboratory where they will be stored at -86 degrees Celsius. The Periopaper samples will be treated for the detection and quantification of the following cytokines: Interleukin-2, Interleukin-4, Interleukin-6, Interleukin-8, Interleukin-10, Tumor Necrosis Factor alpha and Interferon gamma.

Periapicals will be taken at baseline and 12 months. All radiographs will be standardized.

After 12 months, the implant crown will be removed and the implant crown's surface alterations will be evaluated using atomic force microscopy (AFM) using the RA, or average roughness, and the RZ, or mean roughness depth, scores. The implant crown surface will then be repolished/reglazed and delivered back to the patient's mouth. Crowns will be evaluated before delivery to determine adequate level of smoothness.

Based on the presence of cytokines in the Peri-implant Crevicular Fluid, the degree of surface alterations, the modified plaque index, implant probing depths, full mouth plaque index, and full mouth bleeding on probing, we can determine if scratching affects the inflammation around the screw retained dental implant.

ELIGIBILITY:
Inclusion criteria:

* patients who require a single unit implant crown
* patients requiring a single, screw retained, zirconia implant supported crown
* patient who are non-smokers

Exclusion Criteria:

* patients on corticosteroids
* patients who have used antibiotics within the preceding 3 months
* patients with uncontrolled diabetes mellitus
* patients on daily nonsteroidal anti-inflammatory drugs
* patients who are smokers.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Degree of surface roughness | 12 months
  The implant crown's surface alterations will be evaluated using atomic force microscopy (AFM) using the average roughness (Ra) and the mean roughness depth (Rz), scores. Crowns will be evaluated before delivery to determine adequate level of smoothness. For our study, Ra and Rz should range from 0.1µm to 0.5µm. Higher values represent more scratching.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba; College of Dentistry; Faculty of Periodontics, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fugazzotto PA, Gulbransen HJ, Wheeler SL, Lindsay JA. The use of IMZ osseointegrated implants in partially and completely edentulous patients: success and failure rates of 2,023 implant cylinders up to 60+ months in function. Int J Oral Maxillofac Implants. 1993;8(6):617-21. PMID 8181823
- [Background] Lindquist LW, Carlsson GE, Jemt T. A prospective 15-year follow-up study of mandibular fixed prostheses supported by osseointegrated implants. Clinical results and marginal bone loss. Clin Oral Implants Res. 1996 Dec;7(4):329-36. doi: 10.1034/j.1600-0501.1996.070405.x. PMID 9151599
- [Background] Lindh T, Gunne J, Tillberg A, Molin M. A meta-analysis of implants in partial edentulism. Clin Oral Implants Res. 1998 Apr;9(2):80-90. doi: 10.1034/j.1600-0501.1998.090203.x. PMID 9663035
- [Background] Baek SH, Shon WJ, Bae KS, Kum KY, Lee WC, Park YS. Evaluation of the safety and efficiency of novel metallic ultrasonic scaler tip on titanium surfaces. Clin Oral Implants Res. 2012 Nov;23(11):1269-74. doi: 10.1111/j.1600-0501.2011.02302.x. Epub 2011 Sep 30. PMID 22093039
- [Background] Mann M, Parmar D, Walmsley AD, Lea SC. Effect of plastic-covered ultrasonic scalers on titanium implant surfaces. Clin Oral Implants Res. 2012 Jan;23(1):76-82. doi: 10.1111/j.1600-0501.2011.02186.x. Epub 2011 Apr 13. PMID 21488970
- [Background] Fakhravar B, Khocht A, Jefferies SR, Suzuki JB. Probing and scaling instrumentation on implant abutment surfaces: an in vitro study. Implant Dent. 2012 Aug;21(4):311-6. doi: 10.1097/ID.0b013e3182588822. PMID 22814556
- [Background] Park JB, Kim N, Ko Y. Effects of ultrasonic scaler tips and toothbrush on titanium disc surfaces evaluated with confocal microscopy. J Craniofac Surg. 2012 Sep;23(5):1552-8. doi: 10.1097/SCS.0b013e31825e3ba6. PMID 22976659
- [Background] Unursaikhan O, Lee JS, Cha JK, Park JC, Jung UW, Kim CS, Cho KS, Choi SH. Comparative evaluation of roughness of titanium surfaces treated by different hygiene instruments. J Periodontal Implant Sci. 2012 Jun;42(3):88-94. doi: 10.5051/jpis.2012.42.3.88. Epub 2012 Jun 30. PMID 22803010
- [Background] Kawashima H, Sato S, Kishida M, Yagi H, Matsumoto K, Ito K. Treatment of titanium dental implants with three piezoelectric ultrasonic scalers: an in vivo study. J Periodontol. 2007 Sep;78(9):1689-94. doi: 10.1902/jop.2007.060496. PMID 17760537
- [Background] Sato S, Kishida M, Ito K. The comparative effect of ultrasonic scalers on titanium surfaces: an in vitro study. J Periodontol. 2004 Sep;75(9):1269-73. doi: 10.1902/jop.2004.75.9.1269. PMID 15515344
- [Background] Augthun M, Tinschert J, Huber A. In vitro studies on the effect of cleaning methods on different implant surfaces. J Periodontol. 1998 Aug;69(8):857-64. doi: 10.1902/jop.1998.69.8.857. PMID 9736367
- [Background] Hallmon WW, Waldrop TC, Meffert RM, Wade BW. A comparative study of the effects of metallic, nonmetallic, and sonic instrumentation on titanium abutment surfaces. Int J Oral Maxillofac Implants. 1996 Jan-Feb;11(1):96-100. PMID 8820128
- [Background] Brookshire FV, Nagy WW, Dhuru VB, Ziebert GJ, Chada S. The qualitative effects of various types of hygiene instrumentation on commercially pure titanium and titanium alloy implant abutments: an in vitro and scanning electron microscope study. J Prosthet Dent. 1997 Sep;78(3):286-94. doi: 10.1016/s0022-3913(97)70028-3. PMID 9297646
- [Background] Homiak AW, Cook PA, DeBoer J. Effect of hygiene instrumentation on titanium abutments: a scanning electron microscopy study. J Prosthet Dent. 1992 Mar;67(3):364-9. doi: 10.1016/0022-3913(92)90248-9. PMID 1324308
- [Background] Speelman JA, Collaert B, Klinge B. Evaluation of different methods to clean titanium abutments. A scanning electron microscopic study. Clin Oral Implants Res. 1992 Sep;3(3):120-7. doi: 10.1034/j.1600-0501.1992.030304.x. PMID 1290792
- [Background] Pontoriero R, Tonelli MP, Carnevale G, Mombelli A, Nyman SR, Lang NP. Experimentally induced peri-implant mucositis. A clinical study in humans. Clin Oral Implants Res. 1994 Dec;5(4):254-9. doi: 10.1034/j.1600-0501.1994.050409.x. PMID 7640340